CLINICAL TRIAL: NCT04583163
Title: Inter- and Intra-Observer Variability in Transcranial Doppler (TCD) Technique in Neurocritical Care Patients
Brief Title: Variability in Transcranial Doppler Technique in Neuro-Critical Care Patients
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to resource limitations
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0945
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Aneurysm; Stroke; Vasospasm, Cerebral; Subarachnoid Hemorrhage, Aneurysmal; Aneurysmal Subarachnoid Hemorrhage; Cerebral Ischemia
Keywords: Transcranial Doppler; TCD; Interrater Variability; Intrarater Variability; Transcranial Doppler Ultrasound; Neurocritical Care; DCI; Delayed Cerebral Ischemia; MCA; PCA; Mean Flow Velocity
MeSH Terms: conditions — Intracranial Aneurysm; Stroke; Vasospasm, Intracranial; Subarachnoid Hemorrhage; Brain Ischemia | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Neuro-critical Care Patients: Up to 12 subjects will be recruited over a 1 year period. Patients enrolled in the study are recruited from the pool of neuro-critical care patients admitted to the surgical intensive care unit (SICU).
  To meet study inclusion, TransCranial Doppler (TCD) testing will be ordered as part of the standard of care for these patients. The test will not be ordered solely for research purposes. There are no known side effects from the non-invasive measurement of cerebral blood flow using ultrasound.
  Three different TCD technicians will perform triplicate readings on 3 consecutive days on up to 12 patients already undergoing TCD as ordered by their treating team. Standard of care on specific neuro critical care patients (such as cerebral aneurysms) is to undergo daily TCD monitoring to assess for possible vasospasm. Patients will be in the supine position while measurements are obtained. The probe will be placed in the preauricular region of the temporal window.
  Interventions: Diagnostic Test: Transcranial Doppler

INTERVENTIONS:
Diagnostic Test: Transcranial Doppler — Transcranial Doppler is a non-invasive, painless, ultrasound technique that uses high frequency sound waves to measure the rate and direction of blood flow vessels in the brain.
  Other Names: TCD; TCD Ultrasound; Transcranial Doppler Ultrasound; Transcranial Neurovascular Exam; TCD Study; Transcranial Doppler Study

SUMMARY:
This study aims to determine the inter- and intra-variability of Transcranial Doppler (TCD) ultrasound in neuro-critical care patients who are planned for consecutive daily TCD evaluations.

DETAILED DESCRIPTION:
Patients enrolled in the study are recruited from the pool of neuro-critical care patients admitted to the surgical intensive care unit (SICU). When the patients are admitted in the surgical ICU, the study staff will determine eligibility based on the protocol inclusion criteria. Due to the nature of the disease, there is a high likelihood that patients are either unconscious, of limited mental capacity and/or have been intubated therefore when appropriate the legally authorized representative will be utilized to obtain research consent.

To meet study inclusion, transcranial Doppler (TCD) testing will be ordered as part of the standard of care for these patients. The test will not be ordered solely for research purposes. There are no known side effects from the non-invasive measurement of cerebral blood flow using ultrasound

Three different TCD technicians will do triplicate readings on 3 consecutive days on up to 12 patients already undergoing TCD as ordered by their treating team. Standard of care on specific neuro critical care patients (such as cerebral aneurysms) is to undergo daily TCD monitoring to assess for possible vasospasm. Patients will be in the supine position while measurements are obtained. The probe will be placed in the preauricular region of the temporal window

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older
2. Current hospitalization for a neurologic issue and admitted to the surgical intensive care unit.
3. Undergoing daily transcranial Doppler imaging No
4. English speaking patients and/or legally authorized representative (LAR)

Exclusion Criteria:

1. Less than 18 years of age
2. Patient is unable to obtain consent and no LAR is identified to provide consent
3. Non-English speaking patient or LAR
4. Unable to perform the study due to lack of availability of TCD technologists

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Neuro-critical care patients
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Cohn, MD FACS, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Result] Oyama K, Criddle L. Vasospasm after aneurysmal subarachnoid hemorrhage. Crit Care Nurse. 2004 Oct;24(5):58-60, 62, 64-7. PMID 15526491
- [Result] Kumar G, Shahripour RB, Harrigan MR. Vasospasm on transcranial Doppler is predictive of delayed cerebral ischemia in aneurysmal subarachnoid hemorrhage: a systematic review and meta-analysis. J Neurosurg. 2016 May;124(5):1257-64. doi: 10.3171/2015.4.JNS15428. Epub 2015 Oct 23. PMID 26495942
- [Result] Francoeur CL, Mayer SA. Management of delayed cerebral ischemia after subarachnoid hemorrhage. Crit Care. 2016 Oct 14;20(1):277. doi: 10.1186/s13054-016-1447-6. PMID 27737684
- [Result] Carrera E, Schmidt JM, Oddo M, Fernandez L, Claassen J, Seder D, Lee K, Badjatia N, Connolly ES Jr, Mayer SA. Transcranial Doppler for predicting delayed cerebral ischemia after subarachnoid hemorrhage. Neurosurgery. 2009 Aug;65(2):316-23; discussion 323-4. doi: 10.1227/01.NEU.0000349209.69973.88. PMID 19625911
- [Result] Rigamonti A, Ackery A, Baker AJ. Transcranial Doppler monitoring in subarachnoid hemorrhage: a critical tool in critical care. Can J Anaesth. 2008 Feb;55(2):112-23. doi: 10.1007/BF03016323. PMID 18245071
- [Result] Maeda H, Etani H, Handa N, Tagaya M, Oku N, Kim BH, Naka M, Kinoshita N, Nukada T, Fukunaga R, et al. A validation study on the reproducibility of transcranial Doppler velocimetry. Ultrasound Med Biol. 1990;16(1):9-14. doi: 10.1016/0301-5629(90)90080-v. PMID 2181766
- [Result] Baumgartner RW, Mathis J, Sturzenegger M, Mattle HP. A validation study on the intraobserver reproducibility of transcranial color-coded duplex sonography velocity measurements. Ultrasound Med Biol. 1994;20(3):233-7. doi: 10.1016/0301-5629(94)90063-9. PMID 7914715
- [Result] Totaro R, Marini C, Cannarsa C, Prencipe M. Reproducibility of transcranial Dopplersonography: a validation study. Ultrasound Med Biol. 1992;18(2):173-7. doi: 10.1016/0301-5629(92)90128-w. PMID 1580013
- [Result] Shen Q, Stuart J, Venkatesh B, Wallace J, Lipman J. Inter observer variability of the transcranial Doppler ultrasound technique: impact of lack of practice on the accuracy of measurement. J Clin Monit Comput. 1999 May;15(3-4):179-84. doi: 10.1023/a:1009925811965. PMID 12568169
- [Result] Shrout PE, Fleiss JL. Intraclass correlations: uses in assessing rater reliability. Psychol Bull. 1979 Mar;86(2):420-8. doi: 10.1037//0033-2909.86.2.420. PMID 18839484

RESULTS

PARTICIPANT FLOW:
Groups:
- Neuro-critical Care Patients Receiving Transcranial Doppler Imaging: Neuro-critical care patients admitted to the surgical intensive care unit (SICU) receiving Transcranial Doppler Imaging
Period: Overall Study
Arm/Group | Neuro-critical Care Patients Receiving Transcranial Doppler Imaging
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Neuro-critical Care Patients Receiving Transcranial Doppler Imaging: Neuro-critical care patients receiving Transcranial Doppler Imaging in the neurocritical care unit.
Arm/Group | Neuro-critical Care Patients Receiving Transcranial Doppler Imaging
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 51.7 [50 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Determine the Inter-variability of TCD Ultrasound - EDV Measurement
Description: The inter-variability (agreement among 3 TCD technicians) was measured by using the intraclass correlation coefficient (ICC).
  Three technicians took measurements from the same patient at three different visits. The ICC is calculated based on the readings from the same visit of a patient by different technician as the index for the interrater reliability or agreement among the three technicians. Based on the suggestion from Koo and Li (2016), the interpretation of the agreement by using the ICC is defined as: below 0.50 = poor, 0.50-0.75 = moderate, 0.76-0.90 = good, above 090 = excellent.
Time Frame: 3 consecutive days
Population: Readings from all enrolled participants. Only three patients were enrolled, but each patient was measured by three separate technicians at three different visits, hence the 9 readings (for 3 patients) per visit.
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient (ICC)
Units Other Than Participants: Reading
Groups:
- All Participants: There are no groups/arms for the purpose of this study
Arm/Group | All Participants
Number analyzed (Participants) | 3
Number analyzed (Reading) | 9
intraclass correlation coefficient (ICC)
  End Diastolic Velocity (EDV) Visit 1 | 0.986 [0.874 to 1.000]
  EDV Visit 2 | 0.960 [0.715 to 0.999]
  EDV Visit 3 | 0.817 [0.26 to 0.995]

2. Primary Outcome: Determine the Inter-variability of TCD Ultrasound - PFV Measurement
Description: as for outcome 1
Time Frame: 3 consecutive days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient (ICC)
Units Other Than Participants: Readings
Arm/Group | All Participants
Number analyzed (Participants) | 3
Number analyzed (Readings) | 9
intraclass correlation coefficient (ICC)
  Peak Flow Velocity (PFV) Visit 1 | 0.974 [0.809 to 0.999]
  PFV Visit 2 | 0.973 [0.792 to 0.999]
  PFV Visit 3 | 0.918 [0.558 to 0.998]

3. Primary Outcome: Determine the Inter-variability of TCD Ultrasound - Depth Measurement
Description: as for outcome 1
Time Frame: 3 consecutive days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient (ICC)
Units Other Than Participants: Reading
Arm/Group | All Participants
Number analyzed (Participants) | 3
Number analyzed (Reading) | 9
intraclass correlation coefficient (ICC)
  Depth Visit 1 | 0.938 [0.874 to 1.000]
  Depth Visit 2 | 0.013 [-0.426 to 0.930]
  Depth Visit 3 | 0.904 [0.463 to 0.997]

4. Primary Outcome: Determine the Intra-variability of TCD Ultrasound - EDV Measurement
Description: The intra-variability (reliability or consistency within each TCD technician) was measured by using the intraclass correlation coefficient (ICC).
  Three technicians took measurements from the same patient at three different visits. The ICC is calculated for each technician based on the readings from the same patient.
  Based on the suggestion from Koo and Li (2016), the interpretation of the reliability by using the ICC is defined as: below 0.50 = poor, 0.50-0.75 = moderate, 0.76-0.90 = good, above 090 = excellent.
Time Frame: 3 Consecutive Days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient (ICC)
Units Other Than Participants: Reading
Arm/Group | All Participants
Number analyzed (Participants) | 3
Number analyzed (Reading) | 9
intraclass correlation coefficient (ICC)
  End Diastolic Velocity (EDV) by Technician A | 0.979 [0.773 to 0.999]
  EDV by Technician B | 0.989 [0.880 to 1.000]
  EDV by Technician C | 0.960 [0.576 to 0.999]

5. Primary Outcome: Determine the Intra-variability of TCD Ultrasound - PFV Measurement
Description: as for outcome 4
Time Frame: 3 Consecutive Days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient (ICC)
Units Other Than Participants: Reading
Arm/Group | All Participants
Number analyzed (Participants) | 3
Number analyzed (Reading) | 9
intraclass correlation coefficient (ICC)
  Peak Flow Velocity (PFV) by Technician A | 0.985 [0.837 to 1.000]
  PFV by Technician B | 0.982 [0.812 to 1.000]
  PFV by Technician C | 0.963 [0.611 to 0.999]

6. Primary Outcome: Determine the Intra-variability of TCD Ultrasound - Depth Measurment
Description: as for outcome 4
Time Frame: 3 Consecutive Days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Intraclass Correlation Coefficient
Units Other Than Participants: Reading
Arm/Group | All Participants
Number analyzed (Participants) | 3
Number analyzed (Reading) | 9
Intraclass Correlation Coefficient
  Depth by Technician A | -4.154 [-53.884 to 0.869]
  Depth by Technician B | 0.219 [-7.320 to 0.980]
  Depth by Technician C | 0.008 [-9.563 to 0.975]

7. Secondary Outcome: Change in Velocity Prompting Clinical Intervention
Description: Describe the change in velocity that prompts clinical intervention in symptomatic and asymptomatic vasospasm in neuro-critical care patients.
Time Frame: 3 Consecutive Days
Population: Number of patients who had clinical interventions based on the change in velocity observed.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 3
participants | 0

8. Other Pre Specified Outcome: Summary Statistics for Each Measurement
Description: For each Measurement in the following table, the statistics are based on 27 measurements from those 3 subjects (27 values = 3 subjects * 3 visits on 3 consecutive days * 3 technicians)
Time Frame: Across three visits (during 3 consecutive days)
Population: Based on 27 measurements from those 3 subjects (27 values = 3 subjects * 3 visits during 3 consecutive days* 3 technicians)
Measure: Mean (Standard Deviation); unit: cm/sec
Units Other Than Participants: Readings
Groups:
- End Diastolic Velocity (EDV): EDV measured by Transcranial Doppler (TCD) ultrasound. Measured in cm/s.
- Mean Flow Velocity (MFV): MFV measured by Transcranial Doppler (TCD) ultrasound. Measured in cm/s.
- Peak Flow Velocity (PFV): PFV measured by Transcranial Doppler (TCD) Ultrasound. Measured in cm/s.
Arm/Group | End Diastolic Velocity (EDV) | Mean Flow Velocity (MFV) | Peak Flow Velocity (PFV)
Number analyzed (Participants) | 3 | 3 | 3
Number analyzed (Readings) | 27 | 27 | 27
cm/sec | 37.4 (13.7) | 125.68 (29.77) | 100.8 (21.4)

9. Other Pre Specified Outcome: Summary Statistics for Depth
Description: The statistics are based on 27 measurements from those 3 subjects (27 values = 3 subjects * 3 visits on 3 consecutive days * 3 technicians)
Time Frame: Across three visits (during 3 consecutive days)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Reading
Groups:
- DEPTH: Depth measured by Transcranial Doppler (TCD) ultrasound. Measured in mm.
Arm/Group | DEPTH
Number analyzed (Participants) | 3
Number analyzed (Reading) | 27
mm | 6.8 (7.3)

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Neuro-critical Care Patients Receiving Transcranial Doppler Imaging
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
The study was closed before target enrollment was achieved and only three patients were enrolled. No formal analysis was conducted and as a result of the target enrollment not being achieved, no clinical interventions were introduced or changed as a results of these measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT04583163/Prot_SAP_000.pdf